CLINICAL TRIAL: NCT01641120
Title: Assessing Tolerability of Avonex Intramuscular Injections With a 25 Gauge Needle Versus 30 Gauge Needle
Brief Title: Assessing Tolerability of Avonex Intramuscular Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 11-12-002
Record Dates: First submitted 2012-07-06; First posted 2012-07-16 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Intramuscular Injections; Relapsing Remitting
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30 gauge (Experimental): Subjects used a 30 gauge needle for intramuscular injection of Avonex.
  Interventions: Drug: Avonex
- 25 gauge (Experimental): Subjects used a 25 gauge needle for intramuscular injection of Avonex.
  Interventions: Drug: Avonex

INTERVENTIONS:
Drug: Avonex — Intramuscular injection administered using 25 gauge or 30 gauge needle
  Other Names: Interferon beta-1a

SUMMARY:
The purpose of this study is to evaluate patients' views when injecting Avonex intramuscularly.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 - 65 years of age;
* Confirmed diagnosis of Relapsing Remitting Multiple Sclerosis;
* Currently being treated with Avonex® for at least 90 days;
* Using 25 gauge needles for injection of Avonex® for at least 90 days;
* Willing and able to complete study questionnaires; and
* Provided informed consent to participate in this study

Exclusion Criteria:

* Diagnosis of Progressive Multiple Sclerosis;
* History of recent illness or infection;
* History of allergic reaction to Avonex®;
* Any prior usage of a 30 gauge needle for administration of Avonex®;
* Concurrent treatment with other immunomodulating therapies;
* Pregnant or planning on becoming pregnant;
* Nursing mothers; and
* Unable to complete the requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Wade, MD, Principal Investigator — Mandell Center for Multiple Sclerosis
Locations (1):
- The Mandell Center for Multiple Sclerosis, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 25 Gauge or 30 Gauge Needle: Avonex: Intramuscular injection administered using 25 gauge needle weeks 1, 4, and 5 and 30 gauge needle on weeks 2 and 3.
Period: 25 Gauge Needle Weeks 1, 4, 5
Arm/Group | 25 Gauge or 30 Gauge Needle
Started | 20
Completed | 20
Not Completed | 0
Period: 30 Gauge Needle Weeks 2 and 3
Arm/Group | 25 Gauge or 30 Gauge Needle
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Avonex: Intramuscular injection administered using 30 gauge or 25 gauge needle
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 16
  Black | 3
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Visual Analog Scale Score for Pre-injection Anxiety
Description: The primary endpoint of the study was a change in patient self-reported 100 mm (10 cm) Visual Analogue Scale (VAS) score for pre-injection anxiety. VAS scale (min=0- max=100 mm (10cm)) 0= no anxiety; 100 mm (10 cm)=very severe anxiety.
  Data from Weeks 2 and 3 were combined and averaged to obtain a single value as both weeks a 30 gauge needle was used for injection. The 30 gauge needle VAS mean refers to the mean for pre-injection anxiety for that needle size.
  Data from Weeks 4 and 5 were combined and averaged to obtain a single value as both weeks a 25 gauge needle was used for injection. The 25 gauge needle VAS mean refers to the mean for pre-injection anxiety for that needle size.
Time Frame: Weeks 2, 3, 4, 5
Measure: Mean (Standard Deviation); unit: cm
Groups:
- 25 Gauge: Subjects used a 25 gauge needle for intramuscular injection of Avonex on weeks 4 and 5 of the study.
- 30 Gauge: Subjects used a 30 gauge needle for intramuscular injection of Avonex for weeks 2 and 3 of the study.
Arm/Group | 25 Gauge | 30 Gauge
Number analyzed (Participants) | 20 | 20
cm | 1.58 (2.25) | 2.22 (2.73)
Statistical Analysis 1: Comparison: 25 Gauge vs 30 Gauge; Test type: Superiority or Other; p < .05, Wilcoxon Signed Ranks

2. Secondary Outcome: Fear of Injection
Description: Secondary endpoint was assessment of fear of injection based on patient questionnaires completed prior to each injection. The patient will respond to each statement on a scale which ranges from 1 (almost always) to 4 (almost never).
  Data from Weeks 2 and 3 were combined and averaged to obtain a single value as both weeks a 30 gauge needle was used for injection. Mean describes fear of injection for the 30 gauge needle.
  Data from Weeks 4 and 5 were combined and averaged to obtain a single value as both weeks a 25 gauge needle was used for injection. Mean describes fear of injection for the 25 gauge needle.
Time Frame: Weeks 2, 3, 4, 5
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 30 Gauge: Subjects used a 30 gauge needle for intramuscular injection of Avonex on weeks 2 and 3 of the study.
Arm/Group | 25 Gauge | 30 Gauge
Number analyzed (Participants) | 20 | 20
units on a scale | 1.38 (0.509) | 1.41 (0.558)
Statistical Analysis 1: Comparison: 25 Gauge vs 30 Gauge; Test type: Superiority or Other; p = 0.193, Wilcoxon Signed Ranks

3. Primary Outcome: Visual Analog Scale Score for Post-injection Pain
Description: The primary endpoint of the study was a change in patient self-reported 100 mm (10 cm) Visual Analogue Scale (VAS) score for post-injection pain.VAS scale (min=0 - max=100 mm (10 cm)) 0= no pain; 100 mm (10 cm)=very severe pain.
  Data from Weeks 2 and 3 were combined and averaged to obtain a single value as both weeks a 30 gauge needle was used for injection. The 30 gauge needle VAS mean refers to the mean for post-injection pain for that needle size.
  Data from Weeks 4 and 5 were combined and averaged to obtain a single value as both weeks a 25 gauge needle was used for injection. The 25 gauge needle VAS mean refers to the mean for post-injection pain for that needle size.
Time Frame: Weeks 2, 3, 4, 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 25 Gauge | 30 Gauge
Number analyzed (Participants) | 20 | 20
cm | 1.201 (1.22) | 0.764 (0.93)
Statistical Analysis 1: Comparison: 25 Gauge vs 30 Gauge; Test type: Superiority or Other; p = 0.035, Wilcoxon Signed Ranks

4. Secondary Outcome: Perception of Needle
Description: Secondary endpoint was assessment of the perception of the needle based on patient questionnaires completed after each injection. The patient will respond to each statement on a scale which ranges from 1 (strongly agree) to 5 (strongly disagree).
  A total of 6 statements were given to the participant the more strongly the participant agreed with the statement, the more favorably they perceived the needle.
  Data from Weeks 2 and 3 were combined and averaged to obtain a single value as both weeks a 30 gauge needle was used for injection. Mean describes perception of the 30 gauge needle.
  Data from Weeks 4 and 5 were combined and averaged to obtain a single value as both weeks a 25 gauge needle was used for injection. Mean describes perception of the 25 gauge needle.
Time Frame: Weeks 2, 3, 4, 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25 Gauge | 30 Gauge
Number analyzed (Participants) | 20 | 20
units on a scale | 2.58 (0.914) | 1.94 (0.853)
Statistical Analysis 1: Comparison: 25 Gauge vs 30 Gauge; Test type: Superiority or Other; p = .005, Wilcoxon Signed Ranks

ADVERSE EVENTS:
Groups:
- 25 Gauge: The same subjects used a 25 gauge needle for intramuscular injection of Avonex on weeks 4 and 5 of the study.
Arm/Group | 25 Gauge | 30 Gauge
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No